CLINICAL TRIAL: NCT01262261
Title: A Phase 3, Six-Month, Open-Label, Re-Treatment Study of Probuphine in Opioid Addiction
Brief Title: Re-Treatment Study of Probuphine in Opioid Addiction
Status: Completed | Phase: Phase 3 | Type: Interventional
Sponsor: Titan Pharmaceuticals (Industry)
Responsible Party: Sponsor
Allocation: Non-Randomized | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: PRO-811
Record Dates: First submitted 2010-12-15; First posted 2010-12-17 (Estimated); Last update posted 2018-12-31 (Actual); Status verified 2017-06

CONDITIONS: Opioid Dependency
Keywords: opioid dependence; opioid addiction; buprenorphine; implant; methadone; heroin; suboxone; opioid pain medication; opioid withdrawal
MeSH Terms: conditions — Opioid-Related Disorders | interventions — Buprenorphine

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes

ARMS (1):
- Probuphine (Experimental): patients are first inducted on sublingual buprenorphine then switched to 4 Probuphine Implants
  Interventions: Drug: Probuphine (buprenorphine implant)

INTERVENTIONS:
Drug: Probuphine (buprenorphine implant) — Implantable formulation of buprenorphine made of buprenorphine HCl/ethylene vinyl acetate, considered a drug.

SUMMARY:
Probuphine (buprenorphine implant) is an investigational implant placed just below the skin containing buprenorphine (BPN). BPN is an approved treatment for opioid dependence. This is a 6-month, open-label, re-treatment study that will confirm the safety and efficacy of Probuphine in patients who have previously completed the 6-month PRO-806 study with either Probuphine, placebo or sublingual buprenorphine.

ELIGIBILITY:
Inclusion Criteria:

* Subject has voluntarily provided written informed consent prior to conducting any study-related procedures
* Completion of 24 weeks of treatment in PRO-806
* Subject has been deemed appropriate for entry into this extension study by the investigator
* Females of childbearing potential must be willing to use a reliable means of contraception during the entire study.

Exclusion Criteria:

* An aspartate aminotransferase (AST) levels ≥ 3 X the upper limit of normal, alanine aminotransferase (ALT) levels ≥ 3 X the upper limit of normal, total bilirubin ≥ 1.5 X the upper limit of normal, or creatinine ≥ 1.5 X upper limit of normal on the screening laboratory assessments
* A current diagnosis of chronic pain requiring opioids for treatment
* A pregnant or lactating female
* Current use of agents metabolized through Cytochrome P450 3A4 (CYP 3A4) such as azole antifungals (e.g., ketoconazole), macrolide antibiotics (e.g., erythromycin), or protease inhibitors (e.g., ritonavir, indinavir, and saquinavir)
* A history of coagulopathy within the past 90 days, and/or current anti-coagulant therapy such as warfarin
* A significant medical or psychiatric symptoms, cognitive impairment, or other factors which in the opinion of the Investigator would preclude compliance with the protocol, subject safety, adequate cooperation in the study, or obtaining informed consent
* Any current medical conditions such as severe respiratory insufficiency that may prevent the subject from safely participating in study, or any pending legal action that could prohibit participation or compliance in the study

Ages: 18 Years to 65 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 85 (Actual)
Dates: Start 2010-11; Primary Completion 2011-11 (Actual); Study Completion 2011-11 (Actual)

PRIMARY OUTCOMES:
Number of subjects with Adverse Events (AEs) as a measure of safety | 29 weeks
  AEs that occurred after the signing of the informed consent until 4 weeks after the implants have been removed were followed. Serious AEs and AEs that were designated as possibly related to study drug were followed until resolution or stabilization.

SECONDARY OUTCOMES:
Pharmacokinetic analyses through plasma buprenorphine concentration in subjects as a measure of efficacy | 24 weeks
Percent of subjects retained as a measure of efficacy | 24 weeks
Percent of subjects reporting illicit drug use as a measure of efficacy | 24 weeks
Average daily dose of supplemental sublingual buprenorphine as a measure of efficacy | 24 weeks
Mean total score on SOWS as a measure of efficacy | 24 weeks
Mean total score on COWS as a measure of efficacy | 24 weeks
Mean subjective opioid cravings scores as a measure of efficacy | 24 weeks
Mean total score on Beck Depression Inventory (BDI-II) as a measure of efficacy | 24 weeks
Patient-rated opioid use and problems Responder Analysis as a measure of efficacy | 24 weeks
Physician-rated severity of opioid use and symptoms Responder Analysis as a measure of efficacy | 24 weeks
Overall satisfaction with treatment reported on Patient Satisfaction Survey | 24 weeks

CONTACTS AND LOCATIONS:
Overall Officials: Katherine L. Beebe, Ph.D., Principal Investigator — Titan Pharmaceuticals
Locations (18):
- United States (18):
  - David Geffen School of Medicine at UCLA, Los Angeles, California
  - Synergy Clinical Research Center, National City, California
  - North County Clinical Research, Oceanside, California
  - Friends Research Institute, Torrance, California
  - Amit Vijapura, MD, Jacksonville, Florida
  - Operation PAR, Inc. - TC Campus, Largo, Florida
  - Fidelity Clinical Research, Lauderhill, Florida
  - Scientific Clinical Research, Inc., North Miami, Florida
  - BPRU, Behavioral Biology Research Center, Baltimore, Maryland
  - Stanley Street Treatment and Resources, Inc, Fall River, Massachusetts
  - Precise Research Centers, Flowood, Mississippi
  - Psych Care Consultants Research, St Louis, Missouri
  - St. Luke's Roosevelt Hospital Center, New York, New York
  - Duke University Medical Center, Durham, North Carolina
  - University of Pennsylvania, Philadelphia, Pennsylvania
  - Carolina Clinical Trials, Inc., Charleston, South Carolina
  - University of Vermont, Burlington, Vermont
  - Providence Behavioral Health Services, Everett, Washington

REFERENCES:
- [Background] Ling W, Casadonte P, Bigelow G, Kampman KM, Patkar A, Bailey GL, Rosenthal RN, Beebe KL. Buprenorphine implants for treatment of opioid dependence: a randomized controlled trial. JAMA. 2010 Oct 13;304(14):1576-83. doi: 10.1001/jama.2010.1427. PMID 20940383
- [Background] White J, Bell J, Saunders JB, Williamson P, Makowska M, Farquharson A, Beebe KL. Open-label dose-finding trial of buprenorphine implants (Probuphine) for treatment of heroin dependence. Drug Alcohol Depend. 2009 Jul 1;103(1-2):37-43. doi: 10.1016/j.drugalcdep.2009.03.008. Epub 2009 Apr 28. PMID 19403243
- See also: Related Info — http://www.titanpharm.com